CLINICAL TRIAL: NCT05136768
Title: Phase II Clinical Study of Sintilimab Combined With Platinum-based Chemotherapy and SBRT in the First-line Treatment of Limited Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Sintilimab Combined With Chemotherapy and SBRT in Limited Metastatic Head and Neck Squamous Cell Carcinoma (LM-HNSCC)
Acronym: LM-HNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jun-Lin Yi, MD (Unknown)
Responsible Party: Sponsor-Investigator, Jun-Lin Yi, MD, Vice director of Dept. Radiotherapy, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC3100
Record Dates: First submitted 2021-11-16; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Metastases; Immunotherapy; Stereotactic Body Radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis | interventions — sintilimab; Platinum Compounds; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, single center, single arm, phase II clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Sintilimab combined with platinum-based chemotherapy and SBRT
  Interventions: Drug: Sintilimab; Radiation: SBRT; Drug: Platinum based chemotherapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab: 200mg, administered by intravenous infusion on the first day of each cycle, one cycle every 3 weeks (Q3W), with the maximum cycle of 17. Suspension of Sintilimab administration: patients's request, disease progression, researcher-evaluated SAE
  Other Names: Tyvyt®
Radiation: SBRT — At least one metastatic lesion is suitable for SBRT. If applicable, all metastatic lesions were allowed to be irradiated.
  Recommended dose: BED ≥ 80Gy. Dose fractionation is determined as per physician's discretion, generally depending on the location of irradiated lesion and the distance to surrounding OARs.
  Timing of SBRT: After completing at least 2 platinum-containing chemotherapy plus sintilimab treatments, SBRT can be started after assessing that there is no AE ≥ G2.
  Other Names: SABR
Drug: Platinum based chemotherapy — Platinum based single or doublet chemotherapy, one cycle every 3 weeks (Q3W), 4-6 cycles.
  Other Names: chemotherapy

SUMMARY:
To evaluate the safety and efficacy of combination of Sintilimab and SBRT on the basis of platinum-containing chemotherapy as the first-line treatment of limited metastatic head and neck squamous cell carcinoma (LM-HNSCC).

DETAILED DESCRIPTION:
For patients with LM-HNSCC, the conventional first-line treatment is EXTREME regimen dominated systemic therapy. In the recent era, immunotherapy has emerged to be the paramount issue for cancer treatment. A series of high-quality clinical studies demonstrated that immunotherapy (such as PD1 inhibitor) with or without chemotherapy (depending on CPS status) offered significant survival benefits to patients with recurrent or metastatic (R/M) HNSCC and the toxicities were well tolerated, whereas the PFS was still dismal. SBRT is associated with initiating release of tumor antigens, promoting DC activation, activating APCs, priming CD8+ CTLs, leading to the potential of abscopal effect. Therefore, we hypothesized that adding SBRT to Sintilimab (a PD1 inhibitor) and platinum-containing chemotherapy as the first-line treatment may improve the PFS for limited metastatic head and neck squamous cell carcinoma (LM-HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent before implementing any trial-related procedures;
* Male or female, age ≥18 years old;
* Histologically confirmed head and neck squamous cell carcinoma, which was diagnosed as initial stage IVC/M1(synchronous metastatic disease) according to the 8th edition of UICC/AJCC or previously treated head and neck tumor with newly occurred metachronous metastatic disease ;
* Pathological diagnosis of metastasis is not mandatory, but the clinical diagnosis needs to receive consent of MDT;
* The number of metastases is 1-10;
* PD-L1 expression is positive, CPS≥1;
* According to the evaluation criteria for the efficacy of solid tumors (RECIST version 1.1), at least one metastatic lesion is radiologically measurable;
* Newly-diagnosed HNSCC who has not received any treatment previously or HNSCC who has been diagnosed metastases for the first time after treatment;
* For patients who have received platinum-containing chemotherapy in the past, the interval between the new metastasis and the end of the last chemotherapy administration is at least 6 months;
* After a comprehensive radiological examination, at least one extracranial metastatic lesion with a maximum diameter of ≤ 5cm (which can be treated with SBRT);
* ECOG score 0-1 points;
* Sufficient organ function, subjects need to meet the following laboratory indicators: In the past 14 days without using granulocyte colony stimulating factor, the absolute value of neutrophils (ANC) ≥ 1.5x109/L. In the case of no blood transfusion in the past 14 days, platelets ≥100×109/L. In the past 14 days without blood transfusion or using erythropoietin, hemoglobin>9g/dL；Total bilirubin≤1.5×upper limit of normal (ULN); or total bilirubin>ULN but direct bilirubin≤ULN；Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are within ≤2.5×ULN;Serum creatinine ≤1.5×ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥60 ml/min; Good coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN;Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, subjects whose total T3 (or FT3) and FT4 are within the normal range can also be included in the group;The myocardial enzyme spectrum is within the normal range (if the investigator comprehensively judges that the simple laboratory abnormality is not of clinical significance, it is also allowed to be included);
* Expected survival> 1 year;
* At least one lesion is RECIST 1.1 assessable lesion;
* No previous PD1 or PD-L1 inhibitor treatment history;
* Without comorbidities that needs treatment of immunodepressant;
* Male subjects and women of childbearing age must have contraception within 24 weeks from the start of the study to the last time of using the drug.

Exclusion Criteria:

* The primary site is squamous cell carcinoma of the nasopharynx or skin cancer.
* The number of metastases>10;
* Patients who have been diagnosed with other malignant tumors within 5 years before the first administration and have not been cured (excluding radically cured skin basal cell carcinoma, skin squamous epithelial carcinoma, and/or radically resected carcinoma in situ);
* Currently participating in interventional clinical research treatment, or received other research drugs or used research devices within 4 weeks before the first administration;
* Have received the following therapies in the past: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or for another stimulating or synergistic inhibition of T cell receptors (for example, CTLA-4, OX-40, CD137) drug;
* Received systemic treatment with anti-tumor indications Chinese patent medicines or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use to control pleural fluid) within 2 weeks before the first administration;
* An active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, glucocorticoids, or immunosuppressive agents) occurred within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments;
* Administration of systemic steroid (not include nasal spray, inhalation or other local approach) within 7 days before the first administration of Sintilimab or any other ways of immunosuppression;
* Receiving Xenografts or allogeneic hematopoietic stem cell transplantation in the past;
* Allergic to component of research drugs or adjacent;
* HIV infection;
* Untreated active hepatitis B (HBsAg positive and HBV-DNA copy number larger than upper limit of threshold);
* Untreated active hepatitis C (HCV antibody positive and HCV-RNA larger than upper limit of threshold);
* Inoculation with live vaccine within 30 days before the first administration of Sintilimab;
* Women patients in the pregnancy or lactation period;
* With severe or uncontrollable comorbidity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival time (PFS) | Up to 2 years
  PFS is defined as the duration from the starting date of per-protocol treatment to first progression of disease, death or closure of study.

SECONDARY OUTCOMES:
Overall survival time (OS) | Up to 2 years
  OS was calculated from the starting date of per-protocol treatment to death from any cause.
Objective response rate (ORR) | Up to 1 years
  CR + PR rate according to the RECIST version 1.1 guidelines.
Disease control rate (DCR) | Up to 1 years
  CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Duration of disease response (DOR) | Up to 2 years
  The time from the date of first identification of response (CR or PR) to progression/death (P/D).
Time to progression of initial lesions (TPIL) | Up to 2 years
  The time from the first date of per-protocol treatment to progression of baseline lesions or death.
Time to progression of new lesions (TPNL) | Up to 2 years
  The time from the first date of per-protocol treatment to the appearance of new lesion of tumor or death.
Time to progression of non-irradiated lesions (TPNRL) | Up to 2 years
  Duration from the first date of per-protocol treatment to the specific progression of non-irradiated lesion or death.
Adverse events | Up to 2 years
  Adverse event assessment according to NCI CTCAE 5.0, including AE, TEAE, SAE and irAE.

CONTACTS AND LOCATIONS:
Overall Officials: Junlin Yi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahig H, Aubin F, Stagg J, Gologan O, Ballivy O, Bissada E, Nguyen-Tan FP, Soulieres D, Guertin L, Filion E, Christopoulos A, Lambert L, Tehfe M, Ayad T, Charpentier D, Jamal R, Wong P. Phase I/II trial of Durvalumab plus Tremelimumab and stereotactic body radiotherapy for metastatic head and neck carcinoma. BMC Cancer. 2019 Jan 14;19(1):68. doi: 10.1186/s12885-019-5266-4. PMID 30642290
- [Background] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Background] McBride S, Sherman E, Tsai CJ, Baxi S, Aghalar J, Eng J, Zhi WI, McFarland D, Michel LS, Young R, Lefkowitz R, Spielsinger D, Zhang Z, Flynn J, Dunn L, Ho A, Riaz N, Pfister D, Lee N. Randomized Phase II Trial of Nivolumab With Stereotactic Body Radiotherapy Versus Nivolumab Alone in Metastatic Head and Neck Squamous Cell Carcinoma. J Clin Oncol. 2021 Jan 1;39(1):30-37. doi: 10.1200/JCO.20.00290. Epub 2020 Aug 21. PMID 32822275